CLINICAL TRIAL: NCT02242110
Title: Efficacy of a Brief Treatment for Chronic Nightmares Among Trauma-Exposed Persons With Bipolar Disorder
Brief Title: Brief Treatment for Trauma Nightmares in Trauma-exposed Adults With Bipolar Disorder
Acronym: BERRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Joanne Davis, PI, University of Tulsa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TU1457R1
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Nightmares; Post-traumatic Stress Disorder
Keywords: Nightmares; Sleep; PTSD; Exposure, Relaxation, and Rescripting Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nightmare Treatment (Experimental): The nightmare treatment, Exposure, Relaxation, and Rescripting Therapy for Bipolar disorder (ERRT-Bipolar Disorder), is a weekly 5-session treatment aimed at reducing chronic trauma nightmares and sleep disturbances in adults diagnosed with bipolar disorder.
  Interventions: Behavioral: ERRT-Bipolar Disorder

INTERVENTIONS:
Behavioral: ERRT-Bipolar Disorder — The nightmare treatment, called Exposure, Relaxation, and Rescripting Therapy for Bipolar disorder, is a weekly 5-session treatment aimed at reducing chronic trauma nightmares and sleep disturbances in adults diagnosed with bipolar disorder.
  Other Names: ERRT

SUMMARY:
Exposure, relaxation, and rescripting therapy (ERRT) is a promising psychological intervention developed to target trauma-related nightmares and sleep disturbances. Though further evidence is needed, ERRT has shown strong support in reducing the number and intensity of nightmares, as well as improving overall sleep quality in both civilian and veteran samples. This study will assess the efficacy in individuals diagnosed with bipolar disorder.

DETAILED DESCRIPTION:
This pilot study will examine the efficacy of Exposure, Relaxation, & Rescripting Therapy (ERRT) on chronic nightmares in trauma-exposed adults diagnosed with bipolar disorder (B-ERRT), as these individuals have been excluded from past clinical trials. Eligible participants will be assessed prior to starting treatment. B-ERRT will be conducted once a week for approximately five consecutive weeks for approximately two hours per session. Each treatment session focuses on one of the following topics/skills: psychoeducation regarding trauma, nightmares, and sleep disturbances on bipolar disorder, relaxation techniques, exposure to the trauma-nightmare, and relapse prevention. Participants will then be asked to complete two to three follow-up assessments, 1-week, 3-months, and potentially 1-year after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Nightmares at least once per week for the past month
* Formal diagnosis of Bipolar disorder (I or II)
* Exposure to traumatic event (1+ months ago)
* Stable on bipolar medication for at least 2 months

Exclusion Criteria:

* A traumatic event within the last month
* Intellectual disability
* Current or recent mania/hypomania within the last 3 months
* Suicide attempt or hospitalization within the last 3 months
* Current or untreated substance use disorder within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Past Week Nightmare Frequency | Pre, One week, Three Months
  This fill-in-the-blank variable assesses the number of nightmares experienced in the past week (range = 0 - X nightmares) at each assessment (baseline, one week following treatment, and three months following treatment). Higher values indicate more nightmares (worse outcome).

SECONDARY OUTCOMES:
Change in Clinician Administered PTSD Scale Symptoms | Pre, One week, Three Months
  This semi-structured clinical interview assesses severity of each of 30 items

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Davis, PhD, Principal Investigator — University of Tulsa
Locations (1):
- University of Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis JL, Rhudy JL, Pruiksma KE, Byrd P, Williams AE, McCabe KM, Bartley EJ. Physiological predictors of response to exposure, relaxation, and rescripting therapy for chronic nightmares in a randomized clinical trial. J Clin Sleep Med. 2011 Dec 15;7(6):622-31. doi: 10.5664/jcsm.1466. PMID 22171201